CLINICAL TRIAL: NCT02894723
Title: Efficacy of L-arginine Treatment on Blood Pressure Control Patients With Stage 1 Hypertension
Brief Title: L-arginine Treatment in Mild Hypertension
Acronym: LAHN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0216-15-COM2
Record Dates: First submitted 2016-08-15; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension
Keywords: Hypertension,; Nitric Oxide; L-Arginine; Arterial Stiffness; Ambulatory blood pressure measurement
MeSH Terms: conditions — Hypertension | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- l-arginine (Active Comparator): Patients will receive L-arginine 30 ml twice a day for 8 weeks.
  Interventions: Dietary Supplement: L-arginine
- syrup (Placebo Comparator): Patients will receive placebo, 30 ml twice a day for 8 weeks.
  Interventions: Dietary Supplement: syrup

INTERVENTIONS:
Dietary Supplement: L-arginine — 30 ml arginoline contains 5 gr l-arginine
  Other Names: Arginoline
  Arms: l-arginine
Dietary Supplement: syrup — The same bottle of the experimental group, but without l-arginine
  Other Names: placebo
  Arms: syrup

SUMMARY:
Essential Hypertension is characterized by endothelial dysfunction due to reduced nitric oxide (NO) bioavailability. Impairment in nitric oxide-mediated vasodilatation in human brachial, coronary, and renal arteries has been demonstrated in patients with essential hypertension. Administration of L-arginine, a NO substrate yeld controversial results.

The purpose of the present study, double blind and matched for age, sex and body mass index (BMI), is to assess the efficacy of L-arginine treatment on blood pressure (BP) control and arterial stiffness in patients with stage1 hypertension.

DETAILED DESCRIPTION:
Scientific background

Essential Hypertension is characterized by endothelial dysfunction with impaired vasorelaxation.

Reduced nitric oxide bioavailability, which is considered a hallmark of endothelial dysfunction, plays an important role in mediating blood pressure elevation. Accumulating evidence demonstrates a critical role of nitric oxide in blood pressure regulation. Released from the endothelial cells, nitric oxide increases 30,50-cyclic-guanosine monophosphate (cGMP) production and subsequent cGMP-dependent protein kinase (PKG) activation in the underneath vascular smooth muscle cells (VSMCs), resulting in vasodilatation. The investigators and others have shown that inhibition of NO synthesis increase blood pressure in normal pregnant rats and different animal models. In vivo studies confirmed an essential role of nitric oxide in vasorelaxation of large human arteries. Impairment in nitric oxide-mediated vasodilatation in brachial, coronary, and renal arteries has been demonstrated in patients with essential hypertension.

Several mechanisms have been found responsible for nitric oxide deficiency in hypertension. One of them is deficit of the NO substrate, L-arginine. L-arginine transport is impaired in hypertensive and normotensive patients with a genetic background of essential hypertension, and the offspring of essential hypertensive patients are characterized by a reduced response to acetylcholine linked to a defect in the nitric oxide pathway. These data represent the link between L-arginine and the onset of essential hypertension. The Km of endothelial nitric oxide synthase for L-arginine is about 3mmol/l, but the concentration of plasma L-arginine rarely falls below 60mmol/l in pathological conditions. An elevation in asymmetric dimethylarginine (ADMA, an endogenous NO competitive inhibitor) levels may explain this 'L-arginine paradox'. The administration of excess exogenous L-arginine displaces the competitive inhibitor, improves intracellular transport of this amino acid, and restores NO production to physiological levels. In fact L-arginine supplementation improved endothelial dysfunction in hypertension.

Administration of L arginine in humans have not shown uniform blood pressure responses. A meta-analysis published in 2011 was able to find only 11 articles dealing with l-arginine administration and blood pressure. The population studies were heterogeneous. Compared with placebo, oral L-arginine intervention was associated with an average net change ranging from -23.0 to 2.8 mm Hg for SBP and from -11.0 to 1.0 mm Hg for diastolic BP. Most trials showed an intervention-related trend toward BP reductions, but only a few reached statistical significance.

Endothelial dysfunction leads to an increase in arterial stiffness, a known marker that increases cardiovascular morbidity and mortality. Arterial stiffness can be measured by non invasive methodology, e.g.; measuring carotid-femoral pulse wave velocity, augmentation index, aortic pulse pressure and aortic systolic blood pressure.

Whether administration of l-arginine improved arterial stiffness in patients with mild hypertension it is not known.

Arginoline is a dietary supplement that contains L-arginine at a concentration of 5 g/L. It is possible to dilute with water or take chilled. It is produced by Pharmayeda, an Israeli industry.

Clinical observational studies [personal communication] have shown that at a dose of 60 ml\day [10 gr of l-arginine] flow mediated vasodilation improves, suggesting an increase in nitric oxide function.

Methods

Office Blood Pressure (OBP) measurement:

OBP will be measured with a Suntech 247 digital automated device. BP will be determined 3 times at one min. interval each. The mean of the second and third measurements will be noted as the OBP of the visit.

ABPM:

24 hours ABPM will be performed with an Oscar 2 ABPM device of SunTech Medical. The Oscar 2 ABPM device is clinically validated to all 3 internationally recognized protocols (British Heart Society, American Society of Hypertension and the Association for the Advancement of Medical Instrumentation).

Blood pressure is measured in a 20 min. interval at day time and a 30 min. interval at night time. The patients are requested to fill a diary with their activities during the ABPM study, including their subjective evaluation of the sleeping quality.

Measurement of arterial stiffness:

The SphygmoCor X-CEL System (AtCor Medical, Sydney, Australia) will be used.

The system derives (non invasively) the ascending aortic pressure waveform from the brachial waveform using a validated generalised transfer function.

The SphygmoCor X-CEL system measures the carotid-femoral pulse wave velocity (PWV), the speed of the arterial pressure waveform as it travels through the descending aorta to the femoral artery, which is detected from simultaneously measured carotid and femoral arterial pulses.

Design

The study is a matched double blind study with an experimental group and a placebo group. As the number of the groups is small (20 in each group) the patients will be matched according to age, sex and BMI during the recruitment phase, in order to get to comparable groups. The principal investigator is responsible of the matching.

The experimental group will receive arginoline 30 ml twice a day and the placebo group will receive placebo at the same schedule

Visits:

Week -2:

Sign of informed consent

Office BP. Physical examination. BMI.

Blood exams: Hemoglobin (g%), urea (mg%), creatinine (mg%), Natrium (mEq/l), Potassium (mEq/l), alanine transaminase (ALT),Aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), glucose, cholesterol and triglycerides. and lipid profile.

Urine analysis: microalbuminuria (morning spot)

All patients will receive a booklet with detailed information about healthy life style recommendation to lower blood pressure.

Hypertensive patients on monotherapy will stop treatment.

Week 0

ABPM

Measurement of Central aortic blood pressure and arterial stiffness

Blind group allocation (experimental or placebo group).

Week 2

Office BP measurement.

Week 4

Office BP measurement

Week 6

Office BP measurement

Week 8: ABPM, office BP,

Repeat blood and urine exams as detailed at week -2.

Measurement of Central aortic blood pressure and Arterial stiffness

Statistical evaluation

Will be done using the IBM SPSS statistical software. Pi<0.05 is considered significative

ELIGIBILITY:
Inclusion criteria:

* Stage 1 hypertensive patients, with an office Systolic BP between 140-159 mmHg and/or a diastolic BP between 9-99 mmHg , untreated or treated with monotherapy.
* None to two risk factors [smoking, hyperlipidemia, obesity , family history of cardiovascular disease].
* BMI between 25 to 32.
* Twenty for hours ambulatory blood pressure monitor (ABPM) with a mean Systolic BP of 130-149 mmHg and/or a mean Diastolic BP of 80-89 mmHg.

Exclusion criteria:

* Use of any drug that may affect nitric oxide synthesis and/or blood pressure values (nitrates, antihypertensive drugs, non steroidal anti-inflammatory drugs , steroids, pseudoephedrine).
* Diabetes mellitus.
* Renal failure defined as estimated glomerular filtration rate (eGFR) less than 60 ml/min, using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
* A previous diagnosis of ischemic heart disease, Transient ischemic attack (TIA), Stroke or peripheral arterial disease.
* Patients with recurrent herpes and women who are planning pregnancy during the next year.
* Cancer treated with radiotherapy or chemotherapy during the last year.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure, mmHg | baseline [visit 0] to eight weeks
  change in systolic and/or diastolic blood pressure

SECONDARY OUTCOMES:
Central aortic BP, mmHg | baseline (visit 0) to eight weeks
  changes in Central aortic BP values
Pulse pressure (mmHg) | baseline (visit 0] to eight weeks
  changes in central pulse pressure
Augmentation Index (%) | baseline (visit 0] to eight weeks
  changes in augmentation index
carotid femoral pulse wave velocity (m/s) | baseline (visit 0] to eight weeks
  changes in carotid femoral pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Podjarny, MD, Principal Investigator — Clalit Health Services
Locations (1):
- ADAM Institute of High Blood Pressure, Clalit Health Services, Herzliya, Hasharon Area, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanaka Y, Tang G, Takizawa K, Otsuka K, Eghbali M, Song M, Nishimaru K, Shigenobu K, Koike K, Stefani E, Toro L. Kv channels contribute to nitric oxide- and atrial natriuretic peptide-induced relaxation of a rat conduit artery. J Pharmacol Exp Ther. 2006 Apr;317(1):341-54. doi: 10.1124/jpet.105.096115. Epub 2006 Jan 4. PMID 16394199
- [Background] Li Q, Youn JY, Cai H. Mechanisms and consequences of endothelial nitric oxide synthase dysfunction in hypertension. J Hypertens. 2015 Jun;33(6):1128-36. doi: 10.1097/HJH.0000000000000587. PMID 25882860
- [Background] Joannides R, Haefeli WE, Linder L, Richard V, Bakkali EH, Thuillez C, Luscher TF. Nitric oxide is responsible for flow-dependent dilatation of human peripheral conduit arteries in vivo. Circulation. 1995 Mar 1;91(5):1314-9. doi: 10.1161/01.cir.91.5.1314. PMID 7867167
- [Background] Panza JA, Garcia CE, Kilcoyne CM, Quyyumi AA, Cannon RO 3rd. Impaired endothelium-dependent vasodilation in patients with essential hypertension. Evidence that nitric oxide abnormality is not localized to a single signal transduction pathway. Circulation. 1995 Mar 15;91(6):1732-8. doi: 10.1161/01.cir.91.6.1732. PMID 7882481
- [Background] Treasure CB, Klein JL, Vita JA, Manoukian SV, Renwick GH, Selwyn AP, Ganz P, Alexander RW. Hypertension and left ventricular hypertrophy are associated with impaired endothelium-mediated relaxation in human coronary resistance vessels. Circulation. 1993 Jan;87(1):86-93. doi: 10.1161/01.cir.87.1.86. PMID 8419028
- [Background] Higashi Y, Oshima T, Ozono R, Watanabe M, Matsuura H, Kajiyama G. Effects of L-arginine infusion on renal hemodynamics in patients with mild essential hypertension. Hypertension. 1995 Apr;25(4 Pt 2):898-902. doi: 10.1161/01.hyp.25.4.898. PMID 7721451
- [Background] Taddei S, Virdis A, Mattei P, Ghiadoni L, Sudano I, Salvetti A. Defective L-arginine-nitric oxide pathway in offspring of essential hypertensive patients. Circulation. 1996 Sep 15;94(6):1298-303. doi: 10.1161/01.cir.94.6.1298. PMID 8822983
- [Background] Schlaich MP, Parnell MM, Ahlers BA, Finch S, Marshall T, Zhang WZ, Kaye DM. Impaired L-arginine transport and endothelial function in hypertensive and genetically predisposed normotensive subjects. Circulation. 2004 Dec 14;110(24):3680-6. doi: 10.1161/01.CIR.0000149748.79945.52. Epub 2004 Nov 29. PMID 15569830
- [Background] Forstermann U, Sessa WC. Nitric oxide synthases: regulation and function. Eur Heart J. 2012 Apr;33(7):829-37, 837a-837d. doi: 10.1093/eurheartj/ehr304. Epub 2011 Sep 1. PMID 21890489
- [Background] Boger RH. Asymmetric dimethylarginine, an endogenous inhibitor of nitric oxide synthase, explains the "L-arginine paradox" and acts as a novel cardiovascular risk factor. J Nutr. 2004 Oct;134(10 Suppl):2842S-2847S; discussion 2853S. doi: 10.1093/jn/134.10.2842S. PMID 15465797
- [Background] Naseem KM. The role of nitric oxide in cardiovascular diseases. Mol Aspects Med. 2005 Feb-Apr;26(1-2):33-65. doi: 10.1016/j.mam.2004.09.003. Epub 2005 Jan 24. PMID 15722114
- [Background] Hishikawa K, Nakaki T, Suzuki H, Kato R, Saruta T. Role of L-arginine-nitric oxide pathway in hypertension. J Hypertens. 1993 Jun;11(6):639-45. doi: 10.1097/00004872-199306000-00008. PMID 8397243
- [Background] Ast J, Cieslewicz AR, Korzeniowska K, Bogdanski P, Kazmierczak E, Olszewski J, Skoluda A, Jablecka A. Supplementation with L-arginine does not influence arterial blood pressure in healthy people: a randomized, double blind, trial. Eur Rev Med Pharmacol Sci. 2011 Dec;15(12):1375-84. PMID 22288298
- [Background] Ast J, Jablecka A, Bogdanski P, Smolarek I, Krauss H, Chmara E. Evaluation of the antihypertensive effect of L-arginine supplementation in patients with mild hypertension assessed with ambulatory blood pressure monitoring. Med Sci Monit. 2010 May;16(5):CR266-71. PMID 20424555
- [Background] Gui S, Jia J, Niu X, Bai Y, Zou H, Deng J, Zhou R. Arginine supplementation for improving maternal and neonatal outcomes in hypertensive disorder of pregnancy: a systematic review. J Renin Angiotensin Aldosterone Syst. 2014 Mar;15(1):88-96. doi: 10.1177/1470320313475910. Epub 2013 Feb 22. PMID 23435582
- [Background] Gallagher D, Adji A, O'Rourke MF. Validation of the transfer function technique for generating central from peripheral upper limb pressure waveform. Am J Hypertens. 2004 Nov;17(11 Pt 1):1059-67. doi: 10.1016/j.amjhyper.2004.05.027. PMID 15533735
- [Background] Butlin M, Qasem A, Avolio AP. Estimation of central aortic pressure waveform features derived from the brachial cuff volume displacement waveform. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:2591-4. doi: 10.1109/EMBC.2012.6346494. PMID 23366455
- [Result] Davignon J, Ganz P. Role of endothelial dysfunction in atherosclerosis. Circulation. 2004 Jun 15;109(23 Suppl 1):III27-32. doi: 10.1161/01.CIR.0000131515.03336.f8. PMID 15198963
- [Result] Archer SL, Huang JM, Hampl V, Nelson DP, Shultz PJ, Weir EK. Nitric oxide and cGMP cause vasorelaxation by activation of a charybdotoxin-sensitive K channel by cGMP-dependent protein kinase. Proc Natl Acad Sci U S A. 1994 Aug 2;91(16):7583-7. doi: 10.1073/pnas.91.16.7583. PMID 7519783
- [Result] Podjarny E, Ben-Chetrit S, Rathaus M, Korzets Z, Green J, Katz B, Bernheim J. Pregnancy-induced hypertension in rats with adriamycin nephropathy is associated with an inadequate production of nitric oxide. Hypertension. 1997 Apr;29(4):986-91. doi: 10.1161/01.hyp.29.4.986. PMID 9095088